CLINICAL TRIAL: NCT07212374
Title: Impact of Graduation on Child Development in Uganda - Wave 2 (Ancillary/Extension)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Innovations for Poverty Action (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IPA-2025-UG-Wave2; NCT05531812 (IPA-2022-UG) (Registry Identifier: clinicaltrials.gov); AEARCTR-0004080 (Registry Identifier: AEA RCT Registry)
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Child Development; Under Nutrition; School Readiness; Anemia
Keywords: Uganda; ultra-poor graduation; executive function; IDELA; Raven's Progressive Matrices; hemoglobin; HAZ; WHZ
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pure ("Spillover") Control (C2) (No Intervention): Children aged 0-9 years living in host-community households in pure control communities (no Graduation program) from the parent RCT
- Graduation (T1) (Experimental): Children aged 0-9 years living in host-community households assigned to receive the Graduation program in the parent RCT (no new assignment in Wave 2).
  Interventions: Other: Graduation

INTERVENTIONS:
Other: Graduation — "Graduation" is a multifaceted approach that aims to support ultra-poor households in permanently escaping poverty traps. The standard version of Graduation tested in this study includes: a one-time asset transfer; monthly cash transfers; life skills coaching on topics like health and nutrition; technical skills training on topics like financial literacy; and access to savings services.
  Arms: Graduation (T1)

SUMMARY:
This ancillary/extension study ("Wave 2") measures child development and school readiness outcomes among children residing in households within host communities that participated in the Graduation to Resilience (G2R) randomized controlled trial in Uganda (G2R trial: AEARCTR-0004080 [AEA RCT Registry]; Wave 1 child assessments: NCT05531812). No new randomization or intervention assignment occurs in Wave 2; rather, we assess outcomes in children linked to households in communities previously randomized in the parent study.

Wave 2 expands the eligible child age range (0-9 years) and includes age-appropriate outcomes (e.g., IDELA for school readiness; Raven's Progressive Matrices and executive function tasks for older children). We will compare children in households assigned to receive the Graduation program in the parent RCT (T1) to children in pure ("spillover") control households (C2) in host communities. Primary completion is anticipated in October 2025. Pre-analysis plans for Wave 1 and Wave 2 are posted.

DETAILED DESCRIPTION:
Parent RCT & groups: The G2R trial used staged randomization at the community level. In Wave 2 we sample host-community households only, comparing:

T1 (Graduation): households in host communities assigned to receive the Graduation program in the parent trial;

C2 (pure "spillover" control): households in host control communities.

Wave 2 purpose: To measure child development and school readiness outcomes in an expanded age range (0-9 years) using validated, age-appropriate instruments.

Design note: Wave 2 is observational with exposure defined by prior random assignment in the parent RCT; there is no new assignment of interventions in Wave 2.

Documents: The Pre-Analysis Plan (PAP) for this Wave 2 is available under Study Documents and cross-references the PAP from Wave 1 (NCT05531812).

Linkage to parent study: This record is explicitly linked to NCT05531812 and AEARCTR-0004080 [AEA RCT Registry].

ELIGIBILITY:
Inclusion Criteria:

* Child aged 0-9 years at time of Wave 2 assessment.
* Resides in a host-community household within the G2R trial sample
* Caregiver provides informed consent; child provides assent where applicable.

Exclusion Criteria:

* Caregiver declines consent or child declines assent.
* Not resident in the study communities at time of assessment.

Ages: 6 Months to 119 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2100 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Height-for-age z-score (HAZ) | 6 years after the introduction of Graduation
  Based on WHO Growth Standards
Anemia | 6 years after the introduction of Graduation
  Hemoglobin levels captured using HemoCue devices and categorized according to anemia status (<11.5 g/dL)
Forward Digit Span score | 6 years after the introduction of Graduation
  Children are asked to repeated a sequence of numbers. Children who are successful are presented with progressively longer sequences.
Head-Toes-Knees-Shoulders-Revised (HTKS-R) score | 6 years after the introduction of Graduation
  A self-regulation game which taps children's cognitive flexibility, memory, and self-control. Children are presented with instructions and must remember the rules of a game, which require them to: inhibit the more natural response to instructions in favor of the correct, unnatural one; flexibly shift between old and new rules to commands when given, and; regulate their behavior in accordance with all of the above.
Raven's Progressive Matrices Second Edition score | 6 years after the introduction of Graduation
  A direct assessment of fluid intelligence. Children are presented with 36 items and for each item they are asked to identify the missing piece from a set of options that finishes the matrix/picture that is presented.
IDELA total score | 6 years after the introduction of Graduation
  International Development and Early Learning Assessment (IDELA) total score. Direct assessment of children with items across four domains: literacy, numeracy, motor, and socio-emotional.
Caregiver-Reported Early Development Index (CREDI) overall z-score | 6 years after the introduction of Graduation
  Caregivers report on their child's abilities in the domains of cognitive, language, motor, and social-emotional skills.

SECONDARY OUTCOMES:
Diet diversity | 6 years after the introduction of Graduation
  Number of food groups consumed by the child in the previous 24 hours as reported by the caregiver
Caregiver-child interactions | 6 years after the introduction of Graduation
  Number of different types of interactions between caregiver and child in previous 3 days

OTHER OUTCOMES:
Stunting status | 6 years after the introduction of Graduation
  Height-for-age z-score (HAZ) < -2 based on WHO Growth Standards
Weight-for-height z-score (WHZ) | 6 years after the introduction of Graduation
  Based on WHO Growth Standards
Hemoglobin level | 6 years after the introduction of Graduation
  Hemoglobin levels captured using HemoCue devices
IDELA domain scores | 6 years after the introduction of Graduation
  International Development and Early Learning Assessment (IDELA) scores in the domains of literacy, numeracy, motor, and socio-emotional.

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Brune, PhD, Principal Investigator — Northwestern University; Nathanael Goldberg, MPA, Principal Investigator — Innovations for Poverty Action; Dean Karlan, PhD, Principal Investigator — Northwestern University; Christopher Udry, PhD, Principal Investigator — Northwestern University; Peter Rockers, ScD, Principal Investigator — Boston University; Doug Parkerson, MA, Principal Investigator — Innovations for Poverty Action
Locations (1):
- Innovations for Poverty Action Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Study data will be published in a public repository
Supporting Information: Study Protocol
Time Frame: Study data will be published concurrent with the publication of the manuscript describing the study results.
Access Criteria: All interested researchers will be able to access and download study data without restrictions.

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT07212374/SAP_000.pdf